CLINICAL TRIAL: NCT06242574
Title: A Mixed-methods Study to Identify Meaningful Aspects of Health for Adults With Dementia, Their Care Partners and Healthcare Practitioners
Brief Title: Meaningful Aspects of Health for Adults With Dementia, Their Care Partners and Healthcare Practitioners
Acronym: DiME
Status: Withdrawn | Type: Observational
Why Stopped: Submission to EC abandonned
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23-PP-11
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults with Alzheimer's disease and related dementia: 75 patients with ADRD
  Interventions: Other: Survey
- Care partners of Adults with Alzheimer's disease and related dementia: 75 care partners for adults with ADRD
  Interventions: Other: Survey
- Clinicians who treat patients with Alzheimer's disease and related dementia: 25 healthcare practitioners
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Each group will have to complete a questionnaire online, taking about 30 minutes.

SUMMARY:
The aim of this study is to describe, using a non-interventional survey, the relevant aspects of health in adults with ADRD for the patients themselves, their carers and healthcare professionals. Commonalities and differences between these three stakeholders and according to the severity of the dementia will also be studied.

DETAILED DESCRIPTION:
Alzheimer's disease and related disorders (ADRD) are the sixth leading cause of death among adults. Currently, more than 55 million people worldwide are living with the disease, with nearly 10 million new cases each year. ADRD causes significant economic and care burdens for thousands of families and their communities, with over 60% of caregivers developing depressive symptoms. ADRD is ranked among the most costly diseases for society . It is therefore necessary to intervene in order to combat this devastating disease. As recent guidance from the Food and Drug Administration indicates, there is a need to identify areas and mechanisms for real-world change to improve patients' quality of life.

The European Medicines Agency Expert Advisory Group concluded that there was no consensus on validated outcomes in early-stage ADRD and identified the need to fill these gaps.

To demonstrate the utility of any clinical outcome assessment, it's important to link these measures to real-world experiences. And to create this link, research is needed to better understand the meaningful aspects of the health of Alzheimer's patients and their caregivers. In addition, it is important to understand how these MAHs relate to clinicians' perspectives and their approach to assessing disease severity.

Thus, the aim of this study is to describe, using a non-interventional survey, the relevant aspects of health in adults with ADRD for the patients themselves, their carers and healthcare professionals.

Participants with Alzheimer's disease and related dementia and caregivers will be recruited through the Memory Clinic at the Geriatric Hospital in Nice.

Healthcare practitioners working at Centre de Mémoire de Ressources et de Recherche, or outside the Centre , and actively treating a minimum of 10 adults with ADRD, including: neurologists, geriatricians, psychiatrists, neuropsychologists and social workers will be proposed to participate.

All participants will be given a web link to access the survey and will complete it remotely. The survey will take approximately 30 minutes to complete.

ELIGIBILITY:
Adults with Alzheimer's disease and related dementia:

1. ADRD inclusive of the following :

   * Mild dementia due to Alzheimer's disease inclusive of:

     * Mild Cognitive Impairment (MCI),
     * Prodromal Alzheimer's disease,
     * Subjective cognitive impairment,
     * Early onset dementia due to Alzheimer's disease,
     * Mild Alzheimer's Disease
   * Frontotemporal dementia (FTD) - Frontal variant
   * Frontotemporal dementia (FTD) - Primary progressive aphasia
   * Lewy Body dementia (LBD)
   * Vascular dementia
2. Ability to read, understand and express non opposition
3. Aged 50 years or older
4. Patient affiliated to the social security system

Care partners:

1. Unpaid care partners for adults with Alzheimer's disease and related dementia

   ■ A care partner is the primary person who cares for an adult with ADRD, including but not limited to partner, spouse, family member, or significant other of the individual with ADRD. Care partners will be recruited where they care for patients with:
   * Mild dementia due to Alzheimer's disease (inclusive of Mild Cognitive Impairment (MCI), Prodromal Alzheimer's disease, Subjective cognitive impairment, Early onset dementia due to Alzheimer's disease, Mild Alzhiemer's Disease )
   * Moderate to severe dementia due to Alzheimer's disease
   * Frontotemporal dementia (FTD) - Frontal variant
   * Frontotemporal dementia (FTD) - Primary progressive aphasia
   * Lewy Body dementia (LBD)
   * Vascular dementia
2. Delivers at least 10 hours of additional care per week since diagnosis
3. Ability to read, understand and express non opposition
4. Aged 18 years or older
5. Subject affiliated to the social security system

Health-care practitioners

1. Healthcare practitioners actively treating adults with ADRD, including: neurologists, geriatricians, psychiatrists, neuropsychologists and social workers
2. Currently treats a minimum of 10 ADRD patients
3. express non opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with ADRD, their care givers and Health-care practitioners
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the meaningful aspects of health that patients, care partners and clinicians consider most important when considering improvement in the ADRD patient's condition and when considering prevention of decline in the ADRD patient's condition | day 1
  questionnaire specially developed for the study containing a set of MAH ranking exercises and free text response questions
Assessment of the meaningful aspects of health that patients, care partners and clinicians consider most important when considering prevention of decline in the ADRD patient's condition | day1
  questionnaire specially developed for the study containing a set of MAH ranking exercises and free text response questions

CONTACTS AND LOCATIONS:
Locations (1):
- chu de Nice, Nice, France